CLINICAL TRIAL: NCT05597982
Title: How Do Structural Social Determinants of Health Affect AKT-MP and Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI confirmed this study was withdrawn and did not begin locally.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-387 Supplement
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Kidney Diseases; Social Determinants of Health
Keywords: Transplant
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KTFT (Experimental)
  Interventions: Other: Kidney Transplant Fast Track (KTFT)
- PN (Experimental)
  Interventions: Other: Peer Navigation (PN)

INTERVENTIONS:
Other: Kidney Transplant Fast Track (KTFT) — Streamlined KT evaluation involving completion of most or all testing on the same day a patient arrives for their first pre-transplant clinic appointment. Or, a transplant clinic scheduler secures testing within a 4 week period.
  Arms: KTFT
Other: Peer Navigation (PN) — Uses trained, previous KT recipients who meet weekly to monthly with patient participants to provide tailored information and assistance in completing the necessary steps to proceed to transplant.
  Arms: PN

SUMMARY:
Our parent award compares two patient-centered methods to facilitate KT evaluation:

kidney transplant fast track (FT), a streamlined KT evaluation process; and peer navigators (PN), a peer assisted evaluation program that incorporates motivational interviewing. This pragmatic randomized trial uses a comparative effectiveness approach to assess whether FT or PN can help patients overcome barriers to transplant listing. The aims of the parent study are to: (1) compare FT and PN to assess improvements in kidney transplant (KT) related outcomes and cost effectiveness; (2) examine how each approach effects changes in cultural/contextual factors, concerns about, and ambivalence to KT; and (3) develop a framework for widespread implementation of either approach. Recent guidelines encourage using PhenX toolkit measures for kidney-disease research and clinical data reporting, but research to date has been limited by cross sectional or retrospective analyses, and incomplete or missing data on key variables, and show limited clinical application or interventions. In addition to the several PhenX individual social determinants of health (SDOH) already collected for the parent award, we propose to add PhenX structural SDOH, including concentrated poverty, food swamp, race/ethnic segregation, and social vulnerability, to our baseline data collection for all 398 patient participants under the proposed administrative supplement. Also, we will add a third assessment to determine how and whether the intervention affected post-transplant outcomes. We will follow patients via their medical records through receipt of KT to determine time to receive transplant (from time evaluation started), and type of transplant received (living or deceased donor KT). At ~6 months post-KT, participants will complete a third interview to assess KT patient reported outcomes, including health-related quality of life (QOL) and satisfaction with service.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing kidney transplant evaluation at the University of New Mexico
2. Greater than or equal to 18 years of age
3. Mentally competent

Exclusion Criteria:

1. Inclusion across the lifespan - children less than 18 years of age are excluded because all research-related measurements are designed for patients over the age of 18. Children less than 18 years of age have dissimilar decision-making authority as a result of their developmental stage and dependency on adult guardians who must make all their transplant-related decisions, as required by all pediatric transplant centers. The proposed study focuses only on adult transplant patients.
2. Waitlisted or undergoing evaluation at another transplant center
3. Prior kidney transplant
4. Incarcerated patients
5. Pregnant women
6. Active systemic infection
7. Non-skin malignancy or melanoma in the past 2 years
8. Known cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Time to Transplant | Through study completion, an average of 2-3 years
  Time from evaluation initiation to receipt of transplant

SECONDARY OUTCOMES:
Type of transplant received | Through study completion, an average of 2-3 years
  Living or deceased donor kidney transplant received

OTHER OUTCOMES:
Patient Reported Quality of Life using the PROMIS Scale v1.2 Global Health | Through study completion, an average of 2-3 years
  We will use Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.2 Global Health measure to assess quality of life (QOL). It includes items relevant to patients with kidney disease, including overall health, physical limitations, work, pain, energy, and emotional problems. The measure is brief, based on extensive item banks, has been validated in general and CKD populations, and is favored by the International Consortium for Health Outcomes Measurement (ICHOM) CKD Working Group.
Satisfaction with service using the Client Satisfaction Questionnaire | Through study completion, an average of 2-3 years
  Assesses patient reported satisfaction with services received by the transplant clinic team using the Client Satisfaction Questionnaire by Attkisson and colleagues. The measure is brief, and has been used in many clinical populations, along with our previous research CKD and kidney transplant studies.

IPD SHARING:
Plan to Share IPD: No